CLINICAL TRIAL: NCT04384653
Title: An Open-label, Single-dose, Randomized, Two-way, Two-period Crossover Study to Compare the Pharmacokinetics and Bioavailability of a Novel Furosemide Regimen Administered Subcutaneously Versus the Same Dose (80 mg) Administered Intravenously in Subjects With Chronic Heart Failure
Brief Title: Crossover Study to Compare the Pharmacokinetics and Bioavailability of a Novel Furosemide Regimen Administered Subcutaneously vs. the Same Dose Administered Intravenously in Subjects With Chronic Heart Failure
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: SQ Innovation, Inc. (Industry)
Collaborators: Accel Clinical Services (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: SQI-01-01
Record Dates: First submitted 2020-04-30; First posted 2020-05-12 (Actual); Last update posted 2021-09-20 (Actual); Status verified 2021-09

CONDITIONS: Heart Failure
MeSH Terms: conditions — Heart Failure | interventions — Furosemide

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: Yes

ARMS (2):
- Treatment A (Experimental): Furosemide Injection Solution for subcutaneous administration (80 mg) over 5 hours for Treatment Period 1 and IV Furosemide Injection, USP (80 mg) by IV bolus for Treatment Period 2
  Interventions: Drug: Furosemide Injection Solution for subcutaneous administration (80 mg); Drug: Furosemide Injection, USP; Device: Medfusion 3500 (v6) precision infusion pump
- Treatment B (Experimental): IV Furosemide Injection, USP (80 mg) by IV bolus for Treatment Period 1 and Furosemide Injection Solution for subcutaneous administration (80 mg) over 5 hours for Treatment Period 2
  Interventions: Drug: Furosemide Injection Solution for subcutaneous administration (80 mg); Drug: Furosemide Injection, USP; Device: Medfusion 3500 (v6) precision infusion pump

INTERVENTIONS:
Drug: Furosemide Injection Solution for subcutaneous administration (80 mg) — Furosemide Injection Solution for subcutaneous administration (80 mg)
Drug: Furosemide Injection, USP — Furosemide Injection, USP (10 mg/mL), 80 mg by intravenous administration
Device: Medfusion 3500 (v6) precision infusion pump — Furosemide Injection Solution for subcutaneous administration (80 mg)

SUMMARY:
The proposed study aims to compare the pharmacokinetics and bioavailability of intravenous and subcutaneous Furosemide. Although these regimens are not intended to be bioequivalent, they are both expected to achieve therapeutic plasma levels and induce effective diuresis.

The test formulation in this study is a buffered solution, Furosemide Injection Solution at 30 mg/mL at pH 7.4 (range 7.0 to 7.8) and is intended for SC injection according to the instructions in the protocol. A commercial formulation of Furosemide Injection, USP will serve as the reference drug in this study, which will be administered by IV bolus. It contains furosemide 10 mg/mL in solution at alkaline pH of 8.0 to 9.3 and is marketed for IV and IM injection.

The primary objective of the study is to estimate the absolute bioavailability of furosemide administered by subcutaneous infusion compared with an equivalent dose of furosemide administered by IV bolus administration.

DETAILED DESCRIPTION:
This study will be an open-label, single-dose, randomized, two-way, two-period crossover study in 20 adult subjects previously diagnosed with mild to moderate heart failure (New York Health Association [NYHA] class II/III) being treated with oral furosemide therapy at a dose of ≥40 mg/day. Each subject will complete Screening, Admission, Treatment, and Follow-up Phone Call phases. The Screening Phase will be conducted on an outpatient basis between 28 and 3 days prior to admission. Subjects will be instructed to reduce sodium intake (target <2 g sodium/day) starting 3 days prior to each of the clinical research unit (CRU) admissions. Admission (Day -1) consists of CRU admission and final qualification assessments. The Treatment Phase will comprise two crossover periods separated by a 7-day outpatient fluid re-equilibration washout. Subjects will discontinue oral furosemide at least 24 hours prior to administration of study drug for each Crossover Period (e.g., no oral furosemide should be administered after 10pm the night prior to CRU admission). Subjects will be randomly assigned in a 1:1 ratio to 1 of 2 treatment sequences (AB or BA) to receive both subcutaneous furosemide (Treatment A; Test) and IV furosemide (Treatment B; Reference) in Crossover Periods (i.e., subcutaneous followed by IV or vice versa). Subjects will remain domiciled in the CRU for each treatment Period during the Treatment Phase through 24 hours after administration of study drug, after which time they will be discharged from the CRU if safety parameters are acceptable to the Investigator. Oral furosemide therapy will be re-initiated at discharge after Treatment 1 (i.e., during the 7-day fluid re-equilibration washout) and after Treatment 2 (i.e., between discharge and Follow-up Phone Call). The Follow-up Phone Call Phase will occur 7 days (± 1) after discharge from the CRU following Treatment 2, completing subjects' study participation.

ELIGIBILITY:
Inclusion Criteria:

* An Institutional Review Board (IRB)-approved informed consent is signed and dated prior to any study-related activities.
* Male and female subjects ≥18 and ≤ 80 years of age, with body weight <130 kg and body mass index (BMI) <38 kg/m2.
* Females will be non-pregnant, non-lactating, or post-menopausal, or surgically sterile (e.g., tubal ligation, hysterectomy),
* Females of childbearing potential will use TWO of the following forms of contraception: intrauterine device (IUD), IUD with spermicide, female condom with spermicide, contraceptive sponge with spermicide, an intravaginal system, diaphragm with spermicide, cervical cap with spermicide, a male sexual partner who agrees to use a male condom with spermicide, a sterile sexual partner.
* History of at least 3 months treated heart failure (NYHA class II/III) with presence of symptoms of chronic volume overload requiring ongoing treatment with oral furosemide at a dose of ≥40 mg per day for at least 30 days prior to Day -1.
* Agrees to abstain from using alcohol, caffeine-containing products, and tobacco-/nicotine-containing products while in residence at the CRU.
* Able to participate in the study in the opinion of the Investigator.
* Has the ability to understand the requirements of the study and is willing to comply with all study procedures.

Exclusion Criteria:

* Acute Decompensated Heart Failure (ADHF) or recent history of hospitalization for heart failure in the last 4 weeks.
* Worsening of signs or symptoms of heart failure in the two weeks prior to the Screening, or those expected to require IV loop diuretics or inpatient treatment for heart failure during the study.
* Systolic blood pressure (SBP) <90 mmHg.
* Temperature ≥38°C (oral or equivalent) or sepsis or active infection requiring IV anti-microbial treatment.
* Serum sodium <130 mEq/L and serum potassium <3.5 mEq/L.
* Significant other cardiac abnormalities which may interfere with study participation or study assessments.
* Current or planned treatment during the study with any IV therapies, including inotropic agents, vasopressors, levosimendan, nesiritide or analogues; or mechanical support (intraaortic balloon pump, endotracheal intubation, mechanical ventilation, or any ventricular assist device).
* Subject is cachectic.
* Diagnosed with Type I diabetes mellitus or Type II diabetes requiring insulin therapy.
* Presence or need for urinary catheterization, urinary tract abnormality, or disorder interfering with urination.
* Impaired renal function, defined as an estimated glomerular filtration rate (eGFR) on admission <45 mL/min/1.73m2, calculated using the simplified Modification of Diet in Renal Disease (sMDRD) equation.
* Indication of moderate-to-severe hepatic dysfunctions as determined by the Investigator.
* Administration of IV radiographic contrast agent within 72 hours prior to Screening or acute contrast-induced nephropathy at the time of Screening.
* Major surgery within 30 days prior to Screening.
* Administration of an investigational drug or implantation of investigational device, or participation in another interventional trial, within 30 days prior to Screening.
* Any surgical or medical condition, which in the opinion of the Investigator may pose an undue risk to the subject, interfere with participation in the study, or which may affect the integrity of the study data.
* Positive test for hepatitis B (HBsAg), hepatitis C (HCV), or human immunodeficiency virus (HIV) at Screening.
* Any positive urine drug screen at Screening or clinic admission.
* Concomitant use of any drugs known to interact with furosemide.
* History of alcohol abuse within 6 months prior to Screening and/or signs or symptoms of alcoholism, as determined by the Investigator.
* Any positive alcohol test on admission to the CRU.
* History of severe allergic or hypersensitivity reactions to furosemide.
* Donation of greater than 100 mL of either whole blood or plasma within 30 days prior to study drug administration.
* Been informed of possible COVID-19 exposure in past 4 weeks, or recent onset of signs or symptoms of possible COVID-19 infection, including cough, shortness of breath, or temperature ≥ 38°C .
* Traveled via airplane or cruiseship within the last 14 days.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-10-17 (Actual); Primary Completion 2021-06-12 (Actual); Study Completion 2021-06-12 (Actual)

PRIMARY OUTCOMES:
Bioavailability | 0 to 24 hours
  Relative absolute bioavailability following 5-hour subcutaneous infusion based on a comparison of AUC (subcutaneous: IV) of furosemide

SECONDARY OUTCOMES:
Pharmacokinetic parameters | 0 to 24 hours
  PK parameters over the timeframe of 24 hours, including, but not limited to, maximum plasma concentration (Cmax), and time to Cmax (Tmax).
Pharmacokinetic parameters | 0 to 24 hours
  PK parameters over the timeframe of 24 hours, including, but not limited to, area under the concentration versus time curve (AUC) from time 0 (pre-dose) to 24 hours post-dose (AUC0-24), AUC from time 0 to the last measurable plasma concentration (AUClast) and to infinity (AUCinf), half-life (tó), apparent systemic clearance and volume of distribution (subcutaneous only), and systemic clearance and volume of distribution (IV only).
Urine volume | 0 to 24 hours
  Urine volume collected over 8 hours and 24 hours post-dose.
Sodium concentration in urine | 0 to 24 hours
  Sodium concentration in urine collected over 8 hours and 24 hours post-dose.
Pain and discomfort | 0 to 5 hours
  Infusion site pain/discomfort (IV and subcutaneous administration) measured using patient reported scales.
Pain and discomfort | 0 to 5 hours
  Infusion site pain/discomfort (IV and subcutaneous administration) measured using presence of erythema and edema both recorded through photography and assessed by Principal Investigator (PI)/designee-reported scales.

CONTACTS AND LOCATIONS:
Overall Officials: Bruce G Rankin, DO, CPI, FACOFP, Principal Investigator — Accel Research Sites - DeLand Clinical Research Unit
Locations (1):
- Accel Research Sites - DeLand Clinical Research Unit, DeLand, Florida, United States

IPD SHARING:
Plan to Share IPD: No